CLINICAL TRIAL: NCT00607971
Title: A Phase III, Multicenter, Open Label, Extension Study to Evaluate the Long-Term Safety of Renzapride 4 mg Once Daily in Women With Constipation-Predominant Irritable Bowel Syndrome (IBS-C)
Brief Title: Long-Term Safety of Renzapride in Women With Constipation-Predominant Irritable Bowel Syndrome (IBS-C)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to insufficient efficacy over placebo in Study ATL1251/038/CL.
Sponsor: Alizyme (Industry)
Responsible Party: Research & Development Director, Alizyme Therapeutics Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ATL1251/052/CL
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Constipation-Predominant Irritable Bowel Syndrome
Keywords: Constipation predominant irritable bowel syndrome
MeSH Terms: interventions — renzapride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All subjects take two capsules (2x renzapride 2 mg) daily, from the day of enrolment until the scheduled visit at the end of Week 52
  Interventions: Drug: Renzapride

INTERVENTIONS:
Drug: Renzapride — All subjects take two capsules (2x renzapride 2 mg) daily, from the day of enrolment until the scheduled visit at the end of Week 52
  Other Names: ATL-1251; BRL 24924

SUMMARY:
The main purpose of this study is to evaluate the long-term safety and tolerability of renzapride at a dose of 4 mg taken once daily for 12 months in women with constipation-predominant irritable bowel syndrome (IBS-C).

DETAILED DESCRIPTION:
Since IBS is a chronic condition affecting patients over many years, it is anticipated that renzapride will be prescribed and used by patients on a daily basis for long periods of time. Hence the need to understand its long-term safety and tolerability in the target population. This study is open label and so all subjects will take renzapride and will know that they are taking it. Enrolment in to this study is restricted to subjects completing a 12-week, placebo-controlled study of the effectiveness of renzapride in providing relief from IBS-C (Study no. ATL1251/038/CL).

ELIGIBILITY:
Inclusion Criteria:

* completed 12 weeks treatment in the preceding pivotal study ATL1251/038/CL

Exclusion Criteria:

* Subjects who are pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 939 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Adverse events | One year

SECONDARY OUTCOMES:
Vital signs, routine clinical laboratory data, 12-lead ECG | One year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lembo, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Boston
Locations (115):
- United States (115):
  - Research Site, Huntsville, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Sierra Vista, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, North Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site, Carmichael, California
  - Research Site, Cerritos, California
  - Research Site, Chula Vista, California
  - Research Site, Cypress, California
  - Research Site, Laguna Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Carlos, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Lakewood, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Bristol, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pembrook Pines, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Plantation, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Newnan, Georgia
  - Research Site, Rockford, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Arkansas City, Kansas
  - Research Site, Overland Park, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Shreveport, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Laurel, Maryland
  - Research Site, Pasadena, Maryland
  - Research Site, Severna Park, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Chesterfield, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Tupelo, Mississippi
  - Research Site, Mexico, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, Scottsbluff, Nebraska
  - Research Site, Cedar Knolls, New Jersey
  - Research Site, Passaic, New Jersey
  - Research Site, Sicklerville, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Johnson City, New York
  - Research Site, Kingston, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Burlington, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Elkin, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Mogadore, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Downington, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Greer, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Corsicana, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Murray, Utah
  - Research Site, Chesapeake, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Spokane, Washington
  - Research Site, Milwaukee, Wisconsin